CLINICAL TRIAL: NCT06655779
Title: Performance of the Acoustic Based CADScor System in Coronary Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: INTEGRIS Baptist Medical Center (Other)
Responsible Party: Principal Investigator, INTEGRIS Cardiovascular Research, M.D., Medical Director of Cardiology Quality, Informatics and Diagnostic Services., INTEGRIS Baptist Medical Center
Other Study IDs: Integrisbmc
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Angina (stable)
Keywords: CADScore
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Acoustic Detection of Blood Flow — Subject will have the acoustic device scoring performed prior to a Coronary CTA. No treatment decisions will be based upon the acoustic device score.

SUMMARY:
The purpose of this study is to determine if the CAD Score, collected from the CADscore system, performs as well as the Coronary CTA in determining Coronary Artery Disease, in low to intermediate risk patients that are referred for coronary CTA.

ELIGIBILITY:
Inclusion:

* Signed ICF
* Male or female, aged 30 years or above
* Symptoms suggestive of stable coronary artery disease
* No history of coronary artery disease(prior myocardial infarction, percutaneous coronary intervention or coronary artery bypass graft).

Exclusion:

* Asymptomatic for angina or chest pain
* Implanted donor heart
* Previous Coronary Artery Bypass Graft(CABG)
* Previous Coronary Stenting or known CAD
* Arrhythmia causing non-sinus rhythm
* Fragile or compromised skin, or abnormal anatomy or significant operation scars in the fourth left int3er Costal 9IC4-L) recording area
* Implanted mechanical heart or mechanical heart pump
* Implanted pacemaker or Cardioverter Defibrillator(ICD), other implanted active electronics or act5ive electronic support equipment closer than 50 cm to the CADScore System.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects to be recruited from INTEGRIS Baptist Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | From enrollment through 1 year
  To determine that the sensitivity of the CAD score in low to intermediate-risk patients referred for coronary CTA in non-inferior to the device specified sensitivity at 89%.

CONTACTS AND LOCATIONS:
Overall Officials: Jon P Blaschke, MD, Principal Investigator — INTEGRIS Baptist Medical Center
Locations (1):
- INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided